CLINICAL TRIAL: NCT06490029
Title: Evaluation of Hidden Hearing Loss and Vestibular Damage Induced by Anti-cancer Treatments
Brief Title: Diagnostic of Various Ototoxicity Induced by Cancer Treatment
Acronym: BIO-OTOTOX
Status: Recruiting | Type: Observational
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2023RC04
Record Dates: First submitted 2024-06-19; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-06

CONDITIONS: Ototoxicity, Drug-Induced
MeSH Terms: conditions — Ototoxicity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 39 Months
Biospecimen Retention: Samples Without DNA — proteins
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (23):
- A:Previously exposed to CISPLATIN with significant ATL damage: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Previously exposed to CISPLATIN without significant ATL damage: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Previously exposed to cochlear RADIOTHERAPY with significant ATL damage: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Previously exposed to cochlear RADIOTHERAPY WITHOUT significant ATL damage: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Previously exposed to cochlear RADIOTHERAPY & CISPLATIN with significant ATL damage: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Previously exposed to cochlear RADIOTHERAPY & CISPLATIN WITHOUT significant ATL damage: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Previously exposed to OXALIPLATIN: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Previously exposed to CARBOPLATIN: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Previously exposed to TAXANES: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Previously exposed to VINCALCALOIDS: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Previously exposed to other neurotoxicant: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- B:Patients cured of cancer without ototoxic or neurotoxic exposure: Groupe B
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- B:Companions without ototoxic or neurotoxic exposure: Groupe B
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Hyperacusic patients following cancer treatment: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Tinnitus patients following cancer treatment: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- A:Patients with vestibular disorders following cancer treatment: Groupe A
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations
- C:Patients with an indication for CISPLATIN recruited prior to any treatment: Groupe C
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations; Diagnostic Test: Biologic investigations; seric proteins
- C:Patients indicated for cochlear radiotherapy and recruited prior to treatmen: Groupe C
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations; Diagnostic Test: Biologic investigations; seric proteins
- C:Patients with indication for CISPLATIN and cochlear radiotherapy recruited prior any treatment: Groupe C
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations; Diagnostic Test: Biologic investigations; seric proteins
- C:Patients with an indication for OXALIPLATIN treatment recruited prior to any treatment: Groupe C
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations; Diagnostic Test: Biologic investigations; seric proteins
- C:Patients with indication for CARBOPLATIN recruited prior to any treatment: Groupe C
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations; Diagnostic Test: Biologic investigations; seric proteins
- C:Patients with indication for TAXANES therapy recruited prior to any treatment: Groupe C
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations; Diagnostic Test: Biologic investigations; seric proteins
- C:Patients with indication for VINCALCALOIDES or other neurotoxicant: Groupe C
  Interventions: Diagnostic Test: Auditory, vestibular and electrophysiological investigations; Diagnostic Test: Biologic investigations; seric proteins

INTERVENTIONS:
Diagnostic Test: Auditory, vestibular and electrophysiological investigations — otoacoustic emissions, electrocochleography, vocal audiometry in noise and high-frequency tonal audiometry, impedancemetry
Diagnostic Test: Biologic investigations; seric proteins — seric proteins
  Groups: C:Patients indicated for cochlear radiotherapy and recruited prior to treatmen; C:Patients with an indication for CISPLATIN recruited prior to any treatment; C:Patients with an indication for OXALIPLATIN treatment recruited prior to any treatment; C:Patients with indication for CARBOPLATIN recruited prior to any treatment; C:Patients with indication for CISPLATIN and cochlear radiotherapy recruited prior any treatment; C:Patients with indication for TAXANES therapy recruited prior to any treatment; C:Patients with indication for VINCALCALOIDES or other neurotoxicant

SUMMARY:
• Visit the clinic once every 2 weeks for checkups and tests The goal of this clinical trial is to learn if systematic hearing tests (eg fonctional assesment, electrophysiology and seric biomarkers) can diagnose hidden hearing loss or vestibular troubles in a population of patients treated for cancer; population study will include different population in terms of sex/gender, age, medical condition (cancer patients treated with surgery alone and/or radiotherapy and/or chemotherapy, and healthy volunteers).

The main question it aims to answer is:

• To assess the ototoxicity of anticancer drugs using a combination of auditory functional tests (including speech audiometry in noise), vestibular test , plasmatic samples and electrophysiological measures.

Participants will be studied:

Either only after exposition (single visit) Or before, during and after the exposition to potential otototoxic agents with a 4 times Visit the clinic checkups and tests (one before, two while ongoing potential ototoxic agents and 1 post exposition)

Participants will complete questionnaires, undergo audiometric and electrophysiological tests, and their routine biomedical data will be studied, without any modification of the routine care (planned cancer treatment)

DETAILED DESCRIPTION:
Ototoxicity refers to all the auditory and vestibular consequences of a mechanical, radiological and/or chemical aggressor, which can affect these functions via common or specific mechanisms.

Quantification of auditory damage (whatever the type of aggressor) is currently mainly assessed by pure tone audiometry (TTA). However, apart from its subjectivity, LTA only takes into account the audibility of auditory signals - most often only the frequencies of the speech spectrum - and not an individual's ability to analyze and interpret these signals. From an objective point of view, apart from acoustic otoemissions, which have revolutionized neonatal hypoacusis screening, ototoxicity assessment suffers from the absence of reliable biomarkers, objective witnesses of a lesion more or less specific to the type of aggression.

Patients undergoing treatment for cancer are exposed to numerous iatrogenic risks that potentially impact quality of life, whether in a curative or palliative context. In terms of ototoxicity to anticancer drugs (mainly platinum salts), less than half of patients benefit from follow-up during and after exposure to these treatments, despite existing recommendations for cisplatin. There are no recommendations for other anti-cancer drugs (including other platinum salts and neurotoxic drugs) in the absence of clear evidence of a reduction in ATL scores, but the analysis of the literature shows above all a lack of screening for other forms of ototoxicity. Yet the potential consequences of failing to treat hypoacusis can be dramatic: a strong statistical link has been demonstrated, notably with the risk of dementia and mortality, which could also be impacted by the increased risk of falls caused by impaired balance due to vestibulotoxicity (the investigation of which is exceptional in the absence of a vertigo attack).

Areas for improvement include prevention recommendations, improved accessibility to audiometric monitoring, and the development of robust, time-saving diagnostic tests (in patients who often present with other iatrogenic or cancer-induced problems) - the main focus of our study - and the identification of effective treatments.

Vocal noise audiometry (VNA) is an ideal candidate for describing hearing impairment in cancer patients, because :

* Difficulty understanding speech in noise is one of the first signs of hearing loss in the case of peripheral disorders such as presbycusis (linked to ageing) or central auditory disorders, making it possible to account for ototoxicity linked to different mechanisms or damage to different compartments of the auditory system.
* AVB allows assessment under more ecological conditions, i.e., closer to situations encountered in everyday life, than those of tone or voice audiometry in silence, and in a less restrictive way (in terms of time taken to perform the test, and not requiring access to an audiometric booth).

However, the various reference techniques used to assess AVB differ in complexity (comprehension of sentences, syllables, dissyllabic words or logatomes), normative value, conditions and duration, making analysis of intelligibility functions all the more complex. It is generally accepted that logatomes enable us to test the periphery of the auditory system, whereas words and sentences involve mental substitution and the subject's semantic knowledge, and therefore enable us to test hearing in conditions closer to those encountered in everyday life.

In a population particularly exposed to the risk of fatigue and cognitive disorders (chemo-induced cognitive disorders), it is therefore necessary to carry out a study incorporating quality of life questionnaires to take these associated factors into account. In addition, depending on the treatment (and its intensity) and cancer location, different compartments of the auditory system may be affected by the risk of ototoxicity, requiring objective tests (at least on part of our study population) to assess the vestibule, inner ear - in particular to differentiate ciliopathy from cochlear synaptopathy - and middle ear, in order to clarify their respective involvement in functional loss.

The investigators propose to study these parameters in several patient populations, exposed - or not - to ototoxic and/or neurotoxic agents. Comparison within and between these different populations will enable us to assess the specificity and sensitivity of the subjective and objective tests proposed in this study, as well as the validity of composite biomarkers constructed from results on specific groups.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and over
* Registered with social security
* Signed consents
* Absence of presbycusis prior to cancer treatment (groups A and C)
* No known presbycusis (group B)
* Previous exposure to an ototoxic/neurotoxic agent (group A)
* Indication for initiation of ototoxic/neurotoxic therapy (group C)

Exclusion Criteria:

* - Subjects deprived of liberty
* Subjects unable to read or write the French language
* Pregnant and breast-feeding women
* Previous treatment for ototoxicity
* History of bilateral auditory pathology, in particular otosclerosis, perilymphatic fistula, ruptured tympanic membrane, autoimmune hearing loss, acoustic neuroma.
* History of severe head trauma (Glasgow Coma Score <= 8)
* Abnormal otoscopy or tympanometry In addition for group B
* Previous chemotherapy
* Previous ENT radiotherapy
* Ongoing ototoxic drug therapy (quinine, diuretics, aminoglycosides, aspirin, NSAIDs) or corticosteroid therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients treated, not treated or to be treated for cancer or hematologic recquiring neurotoxic treatment
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2024-06-19 (Actual); Primary Completion 2025-03-19 (Estimated); Study Completion 2027-09-19 (Estimated)

PRIMARY OUTCOMES:
Descriptive statistics for audiometry of the various groups | Day 0-Day1 (groups A, B, C) & Day 2, Day 0+7-14-21, Day 0+180-270 (for group C)
  Percentage of correct consonant identification as a function of signal-to-noise ratio for speech audiometry in noise
Descriptive statistics for electrophysiological tests of the various groups | Day 0-Day1 (groups A, B, C) & Day 2, Day 0+7-14-21, Day 0+180-270 (for group C)
  amplitudes of the acoustic distortion products collected during the measurement of induced acoustic otoemissions
Descriptive statistics for protein analyses of the various groups | Day 0-Day1 (groups A, B, C) & Day 2, Day 0+7-14-21, Day 0+180-270 (for group C)
  Concentration of selected proteins in plasma (/mL)

CONTACTS AND LOCATIONS:
Overall Officials: François Régis FERRAND, Study Chair — IRBA, 1 place Valérie André, 91 223 Brétigny-sur-Orge cedex
Locations (1):
- HIA Bégin, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided